CLINICAL TRIAL: NCT02819518
Title: A Randomized, Double-Blind, Phase III Study of Pembrolizumab (MK-3475) Plus Chemotherapy vs Placebo Plus Chemotherapy for Previously Untreated Locally Recurrent Inoperable or Metastatic Triple Negative Breast Cancer - (KEYNOTE-355)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Chemotherapy vs. Placebo Plus Chemotherapy for Previously Untreated Locally Recurrent Inoperable or Metastatic Triple Negative Breast Cancer (MK-3475-355/KEYNOTE-355)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-355; 163422 (Registry Identifier: JAPAN-CTI); MK-3475-355 (Other: MSD); KEYNOTE-355 (Other: MSD); 2016-001432-35 (EudraCT Number)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1: Pembrolizumab + Nab-paclitaxel (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle PLUS nab-paclitaxel 100 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel
- Part 1: Pembrolizumab + Paclitaxel (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel
- Part 1: Pembrolizumab + Gemcitabine/Carboplatin (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS gemcitabine/carboplatin 1000 mg/m^2 (gemcitabine) and an Area Under the Curve (AUC) 2 (carboplatin) on Days 1 and 8 of each 21-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Gemcitabine; Drug: Carboplatin
- Part 2: Pembrolizumab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS one of three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin 1000 mg/m^2 (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin
- Part 2: Placebo + Chemotherapy (Active Comparator): Participants receive placebo (normal saline) IV on Day 1 of each 21-day cycle PLUS one of three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin 1000 mg/m^2 (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin; Drug: Normale Saline Solution

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Part 1: Pembrolizumab + Gemcitabine/Carboplatin; Part 1: Pembrolizumab + Nab-paclitaxel; Part 1: Pembrolizumab + Paclitaxel; Part 2: Pembrolizumab + Chemotherapy
Drug: Nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
  Arms: Part 1: Pembrolizumab + Nab-paclitaxel; Part 2: Pembrolizumab + Chemotherapy; Part 2: Placebo + Chemotherapy
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
  Arms: Part 1: Pembrolizumab + Paclitaxel; Part 2: Pembrolizumab + Chemotherapy; Part 2: Placebo + Chemotherapy
Drug: Gemcitabine — IV infusion
  Other Names: GEMZAR®
  Arms: Part 1: Pembrolizumab + Gemcitabine/Carboplatin; Part 2: Pembrolizumab + Chemotherapy; Part 2: Placebo + Chemotherapy
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
  Arms: Part 1: Pembrolizumab + Gemcitabine/Carboplatin; Part 2: Pembrolizumab + Chemotherapy; Part 2: Placebo + Chemotherapy
Drug: Normale Saline Solution — IV infusion
  Arms: Part 2: Placebo + Chemotherapy

SUMMARY:
The study will consist of two parts.

In Part 1, the safety of pembrolizumab (MK-3475) in combination with one of three different chemotherapies will be assessed in the treatment of locally recurrent inoperable or metastatic triple negative breast cancer (TNBC), which has not been previously treated with chemotherapy.

In Part 2, the safety and efficacy of pembrolizumab plus background chemotherapy will be assessed compared to the safety and efficacy of placebo plus background chemotherapy in the treatment of locally recurrent inoperable or metastatic TNBC, which has not been previously treated with chemotherapy.

The primary hypotheses are that:

1. the combination of pembrolizumab and chemotherapy prolongs Progression-Free Survival (PFS) compared to placebo and chemotherapy in:

   * all participants,
   * participants with programmed cell death-ligand 1 (PD-L1) combined positive score (CPS) ≥1 tumors, and
   * participants with PD-L1 CPS ≥10 tumors, and
2. the combination of pembrolizumab and chemotherapy prolongs Overall Survival (OS) compared to placebo and chemotherapy in:

   * all participants,
   * participants with PD-L1 CPS ≥1 tumors, and
   * participants with PD-L1 CPS ≥10 tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has locally recurrent inoperable breast cancer not previously treated with chemotherapy and which cannot be treated with curative intent OR has metastatic breast cancer not previously treated with chemotherapy.
* Has centrally confirmed TNBC, as defined by the most recent American Society of Clinical Oncology/college of American Pathologists (ASCO/CAP) guidelines.
* Has completed treatment for Stage I-III breast cancer, if indicated, and ≥6 months elapsed between the completion of treatment with curative intent (e.g., date of primary breast tumor surgery or date of last adjuvant chemotherapy administration, whichever occurred last) and first documented local or distant disease recurrence.
* Has been treated with (neo)adjuvant anthracycline, if they received systemic treatment in the (neo)adjuvant setting, unless anthracycline was contraindicated or not considered the best treatment option for the participant in the opinion of the treating physician.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by local radiology review.
* Has provided recently or newly obtained core or excisional biopsy from a locally recurrent inoperable or metastatic tumor lesion for central determination of TNBC status and PD-L1 expression, unless contraindicated due to site inaccessibility and/or participant safety concerns.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 10 days prior to the start of study drug.
* Has a life expectancy ≥12 weeks from randomization.
* Demonstrates adequate organ function, within 10 days prior to the start of study drug.
* Female participants are eligible to participate if they are not pregnant or breastfeeding AND they are not a woman of childbearing potential (WOCBP) OR is a WOCBP using a contraceptive method that is highly effective or is abstinent from heterosexual intercourse during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention AND has a negative highly-sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours (urine) or 72 hours (serum) before the first dose of study intervention.
* Male participants are eligible to participate if they agree to refrain from donating sperm during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention PLUS be abstinent from heterosexual intercourse OR must agree to use contraception unless confirmed to be azoospermic.

Exclusion Criteria:

* Is currently participating in a clinical study and receiving an investigational agent and/or using an investigational device, or has participated in a clinical study and received an investigational agent and/or used an investigational device within 4 weeks prior to randomization.
* Has not recovered (e.g., to ≤ Grade 1 or to baseline) from AEs due to a previously administered therapy.
* Has neuropathy ≥ Grade 2.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (e.g., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.
* Has a known additional malignancy that progressed or required active treatment within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, and in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have stable brain metastases and did not receive chemotherapy for metastatic breast cancer.
* Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has active, or a history of, interstitial lung disease.
* Has a known history of active tuberculosis (TB).
* Has an active infection requiring systemic therapy.
* Has a history of Class II-IV congestive heart failure or myocardial infarction within 6 months of randomization.
* Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days (or longer as specified by local institutional guidelines) after the last dose of study drug.
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T cell receptor (such as cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137) or has previously participated in Merck pembrolizumab (MK-3475) clinical studies.
* Has a known history of human immunodeficiency virus (HIV).
* Has known active hepatitis B or hepatitis C.
* Has received a live vaccine within 30 days prior to randomization.
* Has a known history of hypersensitivity or allergy to pembrolizumab and any of its components and/or to any of the study chemotherapies (e.g., nab-paclitaxel, paclitaxel, gemcitabine, or carboplatin) and any of their components.
* Is receiving any medication prohibited in combination with study chemotherapies as described in the respective product labels, unless medication was stopped within 7 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Im SA, Cortes J, Cescon DW, Yusof MM, Iwata H, Masuda N, Takano T, Huang CS, Chung CF, Tsugawa K, Park YH, Matsumoto K, Inoue K, Kwong A, Loi S, Fu W, Pan W, Karantza V, Rugo HS, Schmid P. Results from the randomized KEYNOTE-355 study of pembrolizumab plus chemotherapy for Asian patients with advanced TNBC. NPJ Breast Cancer. 2024 Sep 12;10(1):79. doi: 10.1038/s41523-024-00679-7. PMID 39266535
- [Derived] Cortes J, Rugo HS, Cescon DW, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Perez-Garcia J, Iwata H, Masuda N, Torregroza Otero M, Gokmen E, Loi S, Guo Z, Zhou X, Karantza V, Pan W, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus Chemotherapy in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2022 Jul 21;387(3):217-226. doi: 10.1056/NEJMoa2202809. PMID 35857659
- [Derived] Cortes J, Cescon DW, Rugo HS, Nowecki Z, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Holgado E, Iwata H, Masuda N, Otero MT, Gokmen E, Loi S, Guo Z, Zhao J, Aktan G, Karantza V, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for previously untreated locally recurrent inoperable or metastatic triple-negative breast cancer (KEYNOTE-355): a randomised, placebo-controlled, double-blind, phase 3 clinical trial. Lancet. 2020 Dec 5;396(10265):1817-1828. doi: 10.1016/S0140-6736(20)32531-9. PMID 33278935
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26179&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants were randomized to Part 1 (Safety Run-in) of the study, and 847 participants were randomized in Part 2 (phase 3) of the study. 12 participants randomized to the Part 2: Pembrolizumab + Chemotherapy arm received a second course of pembrolizumab at the investigator's discretion. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures respectively.
Groups:
- Part 1: Pembrolizumab + Nab-Paclitaxel: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle PLUS nab-paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle.
- Part 1: Pembrolizumab + Paclitaxel: Participants received pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle.
- Part 1: Pembrolizumab + Gemcitabine/Carboplatin: Participants received pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS gemcitabine/carboplatin (gemcitabine) and an Area Under the Curve (AUC) 2 (carboplatin) on Days 1 and 8 of each 21-day cycle.
- Part 2: Pembrolizumab + Chemotherapy: Participants received pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS one of three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle. Qualified participants who received first course of pembrolizumab but continued to experience disease progression were eligible to initiate a second course of pembrolizumab IV Q3W for up to 17 administrations (up to ~1 year).
- Part 2: Placebo + Chemotherapy: Participants received placebo (normal saline) IV on Day 1 of each 21-day cycle PLUS one of three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin 1000 mg/m^2 (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle
Period: Overall Study
Arm/Group | Part 1: Pembrolizumab + Nab-Paclitaxel | Part 1: Pembrolizumab + Paclitaxel | Part 1: Pembrolizumab + Gemcitabine/Carboplatin | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Started | 11 | 14 | 10 | 566 | 281
Treated | 13 (One participant randomized did not receive treatment. 3 participants randomized to Pembrolizumab + Paclitaxel group received Pembrolizumab + Nab-Paclitaxel treatment in error) | 10 (3 participants randomized to Pembrolizumab + Paclitaxel received pembrolizumab + Nab-Paclitaxel in error; 1 participant received pembrolizumab Gemcitabine/Carboplatin in error) | 11 (1 participant randomized to Pembrolizumab + Paclitaxel group received Pembrolizumab + Gemcitabine/Carboplatin in error) | 562 | 281
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 14 | 10 | 566 | 281
Not completed — Death | 9 | 12 | 9 | 475 | 244
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 25 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 1 | 1 | 0 | 34 | 17
Not completed — Transferred to extension study | 1 | 1 | 1 | 32 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Pembrolizumab + Nab-Paclitaxel | Part 1: Pembrolizumab + Paclitaxel | Part 1: Pembrolizumab + Gemcitabine/Carboplatin | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy | Total
Number analyzed (Participants) | 11 | 14 | 10 | 566 | 281 | 882
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (13.5) | 60.4 (15.3) | 59.6 (11.7) | 53.5 (12.7) | 53.0 (12.7) | 53.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 10 | 566 | 281 | 882
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 116 | 48 | 165
  Not Hispanic or Latino | 9 | 14 | 10 | 423 | 218 | 674
  Unknown or Not Reported | 1 | 0 | 0 | 27 | 15 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 11 | 1 | 12
  Asian | 4 | 7 | 4 | 123 | 52 | 190
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 20 | 17 | 38
  White | 6 | 7 | 6 | 384 | 195 | 598
  More than one race | 0 | 0 | 0 | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 17 | 8 | 25
Programmed Cell Death Ligand 1 (PD-L1) Status (Combined Positive Score [CPS] Cutoff of 1) [Count of Participants; unit: Participants] — PD-L1 protein expression in triple-negative breast cancer (TNBC) is determined by using CPS, which is the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100. The number of participants with PD-L1 Status CPS<1 and CPS≥1 at baseline is presented.
  Participants
    PD-L1 CPS ≥1 | 8 | 12 | 7 | 425 | 211 | 663
    PD-L1 CPS <1 | 3 | 2 | 3 | 141 | 70 | 219
PD-L1 Status (CPS Cutoff of 10) [Count of Participants; unit: Participants] — PD-L1 protein expression in TNBC is determined by using CPS, which is the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100. The number of participants with PD-L1 Status CPS<10 and CPS≥10 at baseline is presented.
  Participants
    PD-L1 CPS ≥10 | 1 | 9 | 4 | 220 | 103 | 337
    PD-L1 CPS <10 | 10 | 5 | 6 | 346 | 178 | 545

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Who Experienced an Adverse Event (AE) - All Participants
Description: An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Time Frame: Up to approximately 39 months
Population: All randomly assigned participants who received at least 1 dose of study intervention were included in the group corresponding to the study intervention actually received. Four participants assigned to the pembrolizumab + paclitaxel group received incorrect chemotherapy in error: 3 participants received pembrolizumab + nab-paclitaxel and 1 received pembrolizumab + gemcitabine/carboplatin.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Pembrolizumab + Nab-Paclitaxel | Part 1: Pembrolizumab + Paclitaxel | Part 1: Pembrolizumab + Gemcitabine/Carboplatin
Number analyzed (Participants) | 13 | 10 | 11
Percentage of Participants | 100.0 | 100.0 | 100.0

2. Primary Outcome: Part 1: Percentage of Participants Who Discontinued Study Drug Due to an AE - All Participants
Description: as for outcome 1
Time Frame: Up to approximately 39 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Pembrolizumab + Nab-Paclitaxel | Part 1: Pembrolizumab + Paclitaxel | Part 1: Pembrolizumab + Gemcitabine/Carboplatin
Number analyzed (Participants) | 13 | 10 | 11
Percentage of Participants | 38.5 | 50.0 | 27.3

3. Primary Outcome: Part 2: Progression-Free Survival (PFS) - All Participants
Description: Progression-free survival was defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on assessments by blinded independent central review (BICR) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 53 months
Population: Participants were analyzed in the treatment arm to which they were randomly assigned, regardless of whether they received treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 566 | 281
Months | 7.5 [6.3 to 7.7] | 5.6 [5.4 to 7.2]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0120, Log Rank — One-sided p-value based on log-rank test stratified by chemotherapy (taxane versus [vs] gemcitabine/carboplatin), tumor PD-L1 status (CPS ≥1 vs CPS <1) and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs. no); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.70 to 0.98] — Based on Cox regression model with treatment as a covariate stratified by chemotherapy on study, tumor PD-L1 status, and prior treatment with same class of chemotherapy in the (neo)adjuvant setting

4. Primary Outcome: Part 2: PFS - Participants With Programmed Cell Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1 Tumors
Description: Progression-free survival was defined as the time from randomization to the first documented PD per RECIST 1.1 based on assessments by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 53 months
Population: Participants with PD-L1 CPS ≥1 tumors were analyzed in the treatment arm to which they were randomly assigned, regardless of whether they received treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 425 | 211
Months | 7.6 [6.6 to 8.0] | 5.6 [5.4 to 7.4]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0016, Log Rank — One-sided p-value based on log-rank test stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin), and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs no); Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.62 to 0.91] — Based on Cox regression model with treatment as a covariate stratified by chemotherapy on study, and prior treatment with same class of chemotherapy in the (neo)adjuvant setting

5. Primary Outcome: Part 2: PFS - Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 4
Time Frame: Up to approximately 53 months
Population: Participants with PD-L1 CPS ≥10 tumors were analyzed in the treatment arm to which they were randomly assigned, regardless of whether they received treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 220 | 103
Months | 9.7 [7.6 to 11.3] | 5.6 [5.3 to 7.5]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0018, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.50 to 0.88] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Part 2: Overall Survival (OS) - All Participants
Description: Overall survival is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 53 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 566 | 281
Months | 17.2 [15.3 to 19.0] | 15.5 [13.9 to 17.2]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0797, Log Rank — One-sided p-value based on log-rank test stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin), tumor PD-L1 status (CPS ≥1 vs CPS <1) and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs no); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.76 to 1.05] — [estimate comment as in outcome 3, analysis 1]

7. Primary Outcome: Part 2: OS - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 6
Time Frame: Up to approximately 53 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 425 | 211
Months | 17.6 [15.5 to 19.5] | 16.0 [12.8 to 17.4]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0563, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.04] — [estimate comment as in outcome 4, analysis 1]

8. Primary Outcome: Part 2: OS - Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 6
Time Frame: Up to approximately 53 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 220 | 103
Months | 23.0 [19.0 to 26.3] | 16.1 [12.6 to 18.8]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0093, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.55 to 0.95] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Part 2: Objective Response Rate (ORR) - All Participants
Description: Objective response rate is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experienced a CR or PR as assessed by BICR based on RECIST 1.1 is presented.
Time Frame: Up to approximately 53 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Part 2: Placebo + Chemotherapy: Participants received placebo (normal saline) IV on Day 1 of each 21-day cycle PLUS one three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel 100 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin 1000 mg/m^2 (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle.
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 566 | 281
Percentage of Participants | 40.8 [36.7 to 45.0] | 37.0 [31.4 to 42.9]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.1413, Cochran-Mantel-Haenszel; Difference in ORR (%) vs. Control = 3.8, 95% CI 2-sided [-3.2 to 10.6] — Based on Miettinen & Nurminen method stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin), tumor PD-L1 status (CPS ≥1 vs CPS <1) and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs no)

10. Secondary Outcome: Part 2: ORR - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 9
Time Frame: Up to approximately 53 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 425 | 211
Percentage of Participants | 44.9 [40.1 to 49.8] | 38.9 [32.2 to 45.8]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0725, Cochran-Mantel-Haenszel; Difference in ORR (%) vs. Control = 6.1, 95% CI 2-sided [-2.1 to 14.0] — Based on Miettinen & Nurminen method stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin), and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs no)

11. Secondary Outcome: Part 2: ORR - Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 9
Time Frame: Up to approximately 53 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 220 | 103
Percentage of Participants | 52.7 [45.9 to 59.5] | 40.8 [31.2 to 50.9]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0213, Cochran-Mantel-Haenszel; Difference in ORR(%) vs. Control = 12.1, 95% CI 2-sided [0.4 to 23.4] — Based on Miettinen & Nurminen method stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin) and prior treatment with same class of chemotherapy in the (neo)adjuvant setting (yes vs no)

12. Secondary Outcome: Part 2: Duration of Response (DOR) - All Participants
Description: For participants who demonstrate a confirmed CR (Disappearance of all target lesions) or confirmed PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first, based on assessments by BICR per RECIST 1.1. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 53 months
Population: All randomized participants, regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 231 | 104
Months | NA [NA to NA] — NA indicates median, upper limit, lower limit not reached due to insufficient number of responding participants with relapse | 6.5 [1.5 to NA] — NA indicates upper limit not reached due to insufficient number of responding participants with relapse

13. Secondary Outcome: Part 2: DOR - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 12
Time Frame: Up to approximately 53 months
Population: All randomized participants with PD-LI CPS ≥1 tumors regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 191 | 82
Months | NA [NA to NA] — NA indicates median, upper limit, lower limit not reached due to insufficient number of responding participants with relapse | 6.8 [1.5 to NA] — NA indicates upper limit not reached due to insufficient number of responding participants with relapse

14. Secondary Outcome: Part 2: DOR - Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 12
Time Frame: Up to approximately 53 months
Population: All randomized participants with PD-LI CPS ≥10 tumors regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 116 | 42
Months | NA [NA to NA] — NA indicates median, upper limit, lower limit not reached due to insufficient number of responding participants with relapse | 7.3 [1.5 to NA] — NA indicates upper limit not reached due to insufficient number of responding participants with relapse

15. Secondary Outcome: Part 2: Disease Control Rate (DCR) - All Participants
Description: Disease control rate is defined as the percentage of participants who have achieved CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions) or have demonstrated stable disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]) for at least 24 weeks, based on assessments by BICR per RECIST 1.1.
Time Frame: Up to approximately 53 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 566 | 281
Percentage of Participants | 56.0 [51.8 to 60.1] | 51.2 [45.2 to 57.2]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0966, Cochran-Mantel-Haenszel; Difference in DCR (%) vs. control = 4.7, 95% CI 2-sided [-2.4 to 11.8] — Based on Miettinen & Nurminen method stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin), tumor PD-L1 status (CPS ≥1 vs CPS <1) and prior treatment with same class of chemotherapy in the (neo) adjuvant setting (yes vs no)

16. Secondary Outcome: Part 2: DCR - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 15
Time Frame: Up to approximately 53 months
Population: Participants with PD-L1 CPS ≥1 tumors at baseline were analyzed in the treatment arm to which they were randomly assigned, regardless of whether they received treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 425 | 211
Percentage of Participants | 58.6 [53.7 to 63.3] | 53.6 [46.6 to 60.4]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.1164, Cochran-Mantel-Haenszel; Difference in DCR (%) vs. Control = 5.0, 95% CI 2-sided [-3.2 to 13.1] — Based on Miettinen & Nurminen method stratified by chemotherapy on study (taxane vs gemcitabine/carboplatin) and prior treatment with same class of chemotherapy in the (neo) adjuvant setting (yes vs no)

17. Secondary Outcome: Part 2: DCR - Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 15
Time Frame: Up to approximately 53 months
Population: Participants with PD-L1 CPS ≥10 tumors at baseline were analyzed in the treatment arm to which they were randomly assigned, regardless of whether they received treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 220 | 103
Percentage of Participants | 65.0 [58.3 to 71.3] | 54.4 [44.3 to 64.2]
Statistical Analysis 1: Comparison: Part 2: Pembrolizumab + Chemotherapy vs Part 2: Placebo + Chemotherapy; Test type: Superiority; p = 0.0327, Cochran-Mantel-Haenszel; Difference in DCR (%) vs. Control = 10.8, 95% CI 2-sided [-0.7 to 22.3] — [estimate comment as in outcome 16, analysis 1]

18. Secondary Outcome: Part 2: Percentage of Participants Who Experienced an AE- All Participants
Description: as for outcome 1
Time Frame: Up to approximately 81 months
Population: All randomized participants who received at least 1 dose of study intervention. Participants were included in the group corresponding to the study intervention actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 562 | 281
Percentage of Participants | 98.6 | 98.2

19. Secondary Outcome: Part 2: Percentage of Participants Who Discontinued Study Drug Due to an AE- All Participants
Description: as for outcome 1
Time Frame: Up to approximately 81 months
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 562 | 281
Percentage of Participants | 20.5 | 13.2

20. Secondary Outcome: Part 2: Change From Baseline to Week 15 in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score- All Participants
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" (Item 29) and "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score are presented.
Time Frame: Baseline and Week 15
Population: All randomized participants who received at least 1 dose of study intervention and had completed at least 1 patient-reported outcome (PRO) assessment. Participants were included in the treatment arm to which they were randomly assigned.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 554 | 278
Scores on a scale | -3.52 [-5.61 to -1.42] | -2.15 [-4.97 to 0.67]

21. Secondary Outcome: Part 2: Change From Baseline to Week 15 in EORTC QLQ-C30 Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 20
Time Frame: Baseline and Week 15
Population: All randomized participants with PD-L1 CPS ≥1 tumors who received at least 1 dose of study intervention and had completed at least 1 patient-reported outcome (PRO) assessment. Participants were included in the treatment arm to which they were randomly assigned.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 415 | 208
Scores on a scale | -3.92 [-6.42 to -1.44] | -3.15 [-6.54 to 0.24]

22. Secondary Outcome: Part 2: Change From Baseline to Week 15 in EORTC QLQ-C30 Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score-Participants With PD-L1 CPS ≥10 Tumors
Description: as for outcome 20
Time Frame: Baseline and Week 15
Population: All randomized participants with PD-L1 CPS ≥10 tumors who received at least 1 dose of study intervention and had completed at least 1 patient-reported outcome (PRO) assessment. Participants were included in the treatment arm to which they were randomly assigned.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 216 | 100
Scores on a scale | -2.69 [-5.86 to 0.48] | -0.88 [-5.41 to 3.64]

23. Secondary Outcome: Part 2: Change From Baseline to Week 15 in Systemic Therapy Side Effects Using the EORTC Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23)-All Participants
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and four symptom scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptoms). Participant responses to 7 questions about their systemic therapy side effects were scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score denotes worse symptoms for the systemic therapy side effects symptom scale. The change from baseline in systemic therapy side effects (EORTC QLQ-BR23 Items 1-4, 6, 7, and 8) score is presented.
Time Frame: Baseline and Week 15
Population: as for outcome 20
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 554 | 278
Scores on a scale | 12.50 [10.84 to 14.15] | 12.36 [10.06 to 14.65]

24. Secondary Outcome: Part 2: Change From Baseline to Week 15 in Systemic Therapy Side Effects Using the EORTC QLQ-BR23 - Participants With PD-L1 CPS ≥1 Tumors
Description: as for outcome 23
Time Frame: Baseline and Week 15
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 415 | 208
Scores on a scale | 13.00 [11.08 to 14.91] | 11.86 [9.17 to 14.55]

25. Secondary Outcome: Part 2: Change From Baseline to Week 15 in Systemic Therapy Side Effects Using the EORTC QLQ-BR23- Participants With PD-L1 CPS ≥10 Tumors
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and four symptom scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptoms). Participant responses to 7 questions about their systemic therapy side effects are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score denotes worse symptoms for the systemic therapy side effects symptom scale. The change from baseline in systemic therapy side effects (EORTC QLQ-BR23 Items 1-4, 6, 7, and 8) score is presented.
Time Frame: Baseline and Week 15
Population: as for outcome 22
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part 2: Pembrolizumab + Chemotherapy | Part 2: Placebo + Chemotherapy
Number analyzed (Participants) | 216 | 100
Scores on a scale | 13.56 [10.88 to 16.23] | 13.26 [9.28 to 17.25]

ADVERSE EVENTS:
Time Frame: Up to approximately 81 months
Description: All-cause mortality population: All participants in the treatment arm to which they were randomly assigned. AE population: All participants who received at least 1 dose of study intervention corresponding to the study intervention actually received. 4 participants assigned to the pembrolizumab + paclitaxel group received incorrect chemotherapy in error. Per protocol, "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded..
Groups:
- Part 2: Pembrolizumab + Chemotherapy (First Course): Participants received pembrolizumab 200 mg IV on Day 1 of each 21-day cycle PLUS one of three background chemotherapy regimens at investigator's discretion: 1) nab-paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle, 2) paclitaxel IV on Days 1, 8 and 15 of each 28-day cycle, OR 3) gemcitabine/carboplatin (gemcitabine) and an AUC 2 (carboplatin) on Days 1 and 8 of each 21-day cycle. Qualified participants who received first course of pembrolizumab but continued to experience disease progression were eligible to initiate a second course of pembrolizumab IV Q3W for up to 17 administrations (up to ~1 year).
- Part 2: Pembrolizumab + Chemotherapy (Second Course): Eligible participants received up to 17 additional administrations (up to approximately 1year) of pembrolizumab 200 mg IV on day 1 of each 21-day cycle.
Arm/Group | Part 1: Pembrolizumab + Nab-Paclitaxel | Part 1: Pembrolizumab + Paclitaxel | Part 1: Pembrolizumab + Gemcitabine/Carboplatin | Part 2: Pembrolizumab + Chemotherapy (First Course) | Part 2: Pembrolizumab + Chemotherapy (Second Course) | Part 2: Placebo + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 9/11 | 12/14 | 9/10 | 484/566 | 5/12 | 249/281
Serious Adverse Events (participants affected / at risk) | 3/13 | 4/10 | 9/11 | 169/562 | 3/12 | 68/281
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10 | 11/11 | 551/562 | 11/12 | 273/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Pembrolizumab + Nab-Paclitaxel (N=13) | Part 1: Pembrolizumab + Paclitaxel (N=10) | Part 1: Pembrolizumab + Gemcitabine/Carboplatin (N=11) | Part 2: Pembrolizumab + Chemotherapy (First Course) (N=562) | Part 2: Pembrolizumab + Chemotherapy (Second Course) (N=12) | Part 2: Placebo + Chemotherapy (N=281)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 11 (12) | 0 (0) | 6 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2) | 7 (7) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (14) | 0 (0) | 4 (7)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 6 (7)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fat necrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 4 (6)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 11 (11) | 0 (0) | 7 (7)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Blood corticotrophin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Kidney enlargement (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Assisted suicide (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Pembrolizumab + Nab-Paclitaxel (N=13) | Part 1: Pembrolizumab + Paclitaxel (N=10) | Part 1: Pembrolizumab + Gemcitabine/Carboplatin (N=11) | Part 2: Pembrolizumab + Chemotherapy (First Course) (N=562) | Part 2: Pembrolizumab + Chemotherapy (Second Course) (N=12) | Part 2: Placebo + Chemotherapy (N=281)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 5 (15) | 8 (12) | 294 (633) | 4 (22) | 140 (258)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (64) | 111 (461) | 0 (0) | 50 (158)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 30 (62) | 0 (0) | 4 (15)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (21) | 7 (90) | 232 (936) | 2 (4) | 109 (384)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (89) | 110 (346) | 0 (0) | 56 (155)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (11) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 20 (22) | 0 (0) | 12 (13)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 2 (3) | 1 (1) | 25 (25) | 0 (0) | 4 (4)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (3) | 4 (5) | 85 (96) | 0 (0) | 9 (10)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 20 (20) | 0 (0) | 8 (8)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 6 (6)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (11) | 0 (0) | 8 (8)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (13) | 0 (0) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (6) | 43 (57) | 0 (0) | 25 (28)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 45 (64) | 1 (1) | 16 (19)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (9) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 6 (10) | 155 (212) | 0 (0) | 77 (97)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 2 (3) | 6 (6) | 155 (305) | 1 (2) | 66 (134)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 22 (23) | 0 (0) | 10 (14)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 38 (45) | 0 (0) | 16 (19)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (13) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 18 (18) | 1 (3) | 7 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 15 (16) | 0 (0) | 11 (12)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 2 (3) | 4 (9) | 251 (522) | 1 (1) | 130 (254)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 54 (76) | 0 (0) | 19 (22)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2) | 6 (8) | 140 (248) | 0 (0) | 62 (107)
Asthenia (General disorders) | 6 (16) | 3 (8) | 3 (6) | 108 (194) | 0 (0) | 47 (84)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 25 (27) | 0 (0) | 17 (20)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 16 (18) | 1 (1) | 7 (7)
Fatigue (General disorders) | 1 (1) | 2 (3) | 1 (1) | 180 (258) | 1 (1) | 96 (119)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (3) | 25 (38) | 0 (0) | 14 (25)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 31 (41) | 0 (0) | 14 (21)
Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 0 (0) | 0 (0) | 65 (83) | 0 (0) | 29 (42)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 2 (5) | 99 (150) | 2 (2) | 55 (85)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 3 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 3 (3)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 8 (9) | 1 (2) | 8 (16)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 4 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 7 (9) | 1 (1) | 3 (13)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 11 (13) | 1 (1) | 3 (5)
Erythema infectiosum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 5 (6)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 28 (30) | 0 (0) | 8 (10)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 53 (76) | 1 (1) | 21 (28)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 4 (6)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 0 (0) | 5 (8)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 6 (8)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 4 (4)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (4) | 1 (9) | 58 (94) | 0 (0) | 26 (36)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 49 (70) | 1 (1) | 13 (14)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 9 (14) | 1 (1) | 4 (6)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 0 (0) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 2 (28) | 139 (242) | 2 (2) | 55 (84)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 2 (17) | 131 (225) | 1 (1) | 46 (69)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 50 (79) | 1 (1) | 22 (28)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
Blood corticotrophin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 31 (34) | 0 (0) | 16 (17)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 3 (3)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 20 (35) | 0 (0) | 8 (11)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 14 (19) | 0 (0) | 3 (4)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (7) | 1 (1) | 30 (88) | 2 (17) | 11 (32)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 0 (0) | 1 (38) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (17) | 1 (1) | 128 (668) | 4 (29) | 76 (310)
Neutrophil percentage decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 6 (24) | 0 (0) | 1 (9)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 87 (350) | 2 (10) | 44 (125)
Weight decreased (Investigations) | 1 (2) | 4 (5) | 1 (1) | 50 (55) | 0 (0) | 12 (13)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 14 (14) | 0 (0) | 7 (8)
White blood cell count decreased (Investigations) | 0 (0) | 5 (20) | 2 (3) | 106 (502) | 4 (29) | 55 (211)
Decreased appetite (Metabolism and nutrition disorders) | 8 (12) | 2 (2) | 2 (4) | 118 (140) | 0 (0) | 39 (49)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4) | 27 (40) | 1 (1) | 11 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (48) | 9 (13) | 0 (0) | 8 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (28) | 18 (28) | 0 (0) | 11 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (2) | 28 (46) | 1 (1) | 14 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 15 (23) | 1 (1) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 12 (14) | 0 (0) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (3) | 122 (203) | 0 (0) | 48 (73)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 72 (88) | 1 (2) | 41 (48)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 22 (25) | 0 (0) | 17 (21)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 28 (31) | 0 (0) | 13 (16)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (3) | 59 (83) | 0 (0) | 34 (57)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 25 (28) | 0 (0) | 20 (23)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 56 (68) | 1 (1) | 41 (47)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 10 (11) | 0 (0) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0) | 52 (61) | 0 (0) | 24 (33)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 54 (63) | 0 (0) | 15 (18)
Headache (Nervous system disorders) | 2 (3) | 5 (7) | 1 (1) | 111 (184) | 1 (1) | 66 (104)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 11 (15) | 0 (0) | 3 (5)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (6) | 2 (2) | 1 (1) | 62 (72) | 0 (0) | 35 (50)
Neurotoxicity (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0) | 4 (7) | 0 (0) | 4 (7)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 24 (31) | 0 (0) | 15 (15)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2) | 49 (55) | 0 (0) | 20 (22)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 12 (12) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 4 (5)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 6 (8)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (4) | 23 (23) | 0 (0) | 11 (11)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 20 (20) | 0 (0) | 13 (13)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2) | 2 (2) | 48 (53) | 0 (0) | 28 (32)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 12 (12) | 0 (0) | 3 (3)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (4)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 24 (29) | 0 (0) | 14 (14)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 118 (154) | 0 (0) | 49 (60)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 22 (23) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 69 (82) | 0 (0) | 37 (44)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 20 (26) | 0 (0) | 17 (20)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 29 (32) | 0 (0) | 18 (25)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 12 (12) | 0 (0) | 13 (15)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 2 (2) | 190 (194) | 0 (0) | 97 (97)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 11 (11) | 0 (0) | 6 (7)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 16 (18) | 0 (0) | 10 (10)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 23 (25) | 0 (0) | 11 (18)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 4 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 10 (10)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (6) | 1 (1) | 85 (120) | 1 (1) | 32 (39)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4) | 3 (4) | 110 (154) | 0 (0) | 34 (44)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 25 (41) | 0 (0) | 10 (10)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 0 (0) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 4 (4)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 11 (15) | 0 (0) | 3 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 11 (22) | 0 (0) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 21 (22) | 0 (0) | 10 (14)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 11 (11) | 0 (0) | 9 (10)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 16 (17) | 0 (0) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (2):
  • Study Protocol (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02819518/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02819518/SAP_001.pdf